CLINICAL TRIAL: NCT02976532
Title: Controlling Femoral Derotation Osteotomy With Electromagnetic Tracking - an in Vivo Study
Brief Title: Controlling Femoral Derotation Osteotomy With Electromagnetic Tracking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Dreher, Principal Investigator, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NavDo2014
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Interna Rotation Gait; Cerebral Palsy; Malrotation; Bone; In-toing
Keywords: Electromagnetic tracking; Internal rotation gait; Femoral derotation osteotomy
MeSH Terms: conditions — Cerebral Palsy; Volvulus Of Midgut

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EMT Arm (Other): The study is performed with a single arm, as the system is an additional tool for derotation measurement and the surgical procedure itself and its technique is not changed.
  Interventions: Other: Electromagnetic tracking unit in femoral derotation surgery

INTERVENTIONS:
Other: Electromagnetic tracking unit in femoral derotation surgery — Use of the electromagnetic tracking system during the surgical procedure in addition to the normal measurement with goniometer, the different devices listed are combined to form the EMT system unit
  Other Names: A self developed software interface; EMT pointer device (FlexPointer E01 2002, fiagon GmbH, Berlin, Germany) for surface sampling; EMT sensors embedded in a clamp shell (PointerShell E01 2902, fiagon GmbH, Berlin, Germany); A field generator (AURORA v.2, Northern Digital, Waterloo, Canada)

SUMMARY:
The study is designed to evaluate the use of electromagnetic tracking in femoral derotation osteotomies. The goal is to raise the precision of the surgical procedure in order to improve the outcome in short- and long term. The electromagnetic tracking system is evaluated against a base line CT scan serving as reference standard.

DETAILED DESCRIPTION:
Internal rotation gait is a common deformity in children, especially in those with spastic diplegia. The treatment includes soft tissue and bony correction. Especially the bony procedures e.g. femoral derotation osteotomies have proven to be effective both in short term and long term evaluation. Nonetheless there is still a relevant number of patients that suffer from over- or under-correction and recurrence over time. The reasons are diverse and include false measurement of the derotation in OR.

The study now evaluates electromagnetic tracking for femoral derotation to improve these results.

The patients are recruited from the outpatients department and included if they meet the criteria.

A baseline rotational CT scan and a 3-D-gait analysis are performed and the derotation measured with the EMT system in OR. The results of the measurement is invisible and unknown to the surgeon as the system unit is controlled by a technician.

The surgical procedure follows standard rules and does not need alterations because of the study.

After the operation a second rotational CT scan is performed and the derotation precisely evaluated by two raters and later compared to the results of the electromagnetic tracking system.

ELIGIBILITY:
Inclusion Criteria:

* functionally impairing internal rotation gait and indication for supracondylar derotation osteotomy (Evidence of falling because of internal rotation gait, abnormally increased femoral anteversion, confirmation of internal rotation gait in gait kinematics of hip rotation and foot progression angle and a mid point shift in the clinical examination).

Exclusion Criteria:

* severe mental retardation and inability to undertake the CT scan

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Difference between CT reference measurement and EMT measurement of femoral derotation osteotomies in degrees | After the postoperative CT Scan (maximum of three month after surgery)
  The study evaluates the result of the derotation measurement by the EMT system against the derotation in degrees that is measured with the difference between the pre- and the post-operative CT scan (meaning: EMT measurement intra-operative versus difference in femoral rotation in the CT scan between pre- and post-operative CT). The outcome is given in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dreher, Dr., Principal Investigator — MD
Locations (1):
- Orthopaedic Department, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geisbusch A, Auer C, Dickhaus H, Niklasch M, Dreher T. Electromagnetic bone segment tracking to control femoral derotation osteotomy-A saw bone study. J Orthop Res. 2017 May;35(5):1106-1112. doi: 10.1002/jor.23348. Epub 2016 Jul 4. PMID 27325569